CLINICAL TRIAL: NCT00000563
Title: Prevention of Neonatal Respiratory Distress Syndrome With Antenatal Steroid Administration
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: 201
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Lung Diseases; Respiratory Distress Syndrome
MeSH Terms: conditions — Lung Diseases; Respiratory Distress Syndrome | interventions — Dexamethasone

INTERVENTIONS:
Drug: dexamethasone

SUMMARY:
To determine the effect of corticosteroids, administered 24 to 48 hours before parturition, on the incidence of neonatal respiratory distress syndrome (RDS) and to determine whether the therapy has any adverse short- or long-term (up to 36 months) effects on the infant. Secondarily, to determine whether the therapy has any adverse short-term effects on the mother and to determine whether morbidity rates for neonatal respiratory distress syndrome as well as total and cause-specific infant mortality rates differ between mothers who received antenatal steroids and those who received conventional medical care.

DETAILED DESCRIPTION:
BACKGROUND:

Neonatal respiratory distress syndrome is one of the leading causes of disability and death in the newborn. In the United States, approximately 10 percent of all infants are premature, and each year about 50,000 cases of neonatal respiratory distress syndrome occur.

Extensive studies in animal models on respiratory distress syndrome have demonstrated that antenatal administration of synthetic (dexamethasone) and natural (cortisol) corticosteroids accelerates lung maturation and significantly diminishes the occurrence of RDS. Although a variety of conditions in newborn infants have been treated with steroids over the past 20 years without adverse effects, investigations have been needed on the short-term effects of corticosteroids administered antenatally on neonate and mother and on the long-term effects on the infant.

The Planning Phase of this trial was completed in March 1977, with formulation of a common protocol and manual of operations. Patient screening and enrollment began in August 1977 and ended on March 1, 1980. Follow-up ended in August 1983 and data analysis was completed October 31, 1983.

DESIGN NARRATIVE:

Randomized, double-blind, fixed sample. Six hundred and ninety-six pregnant women were randomized to four doses of dexamethasone every 12 hours or to placebo. Endpoints were the incidence of respiratory distress syndrome and abnormality of motor-neuro-intellectual development in their infants.

ELIGIBILITY:
Male and female fetuses and infants; pregnant women with anticipated premature delivery and gestational age between 26 and 37 weeks.

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1976-06; Study Completion 1983-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Bauer — University of Miami; Richard Depp — Northwestern University; Sheldon Korones — University of Tennessee; Henrique Rigatto — University of Manitoba; Richard Zachman — University of Wisconsin, Madison

REFERENCES:
- [Background] Effect of antenatal dexamethasone administration on the prevention of respiratory distress syndrome. Am J Obstet Gynecol. 1981 Oct 1;141(3):276-87. PMID 7025638
- [Background] Effects of antenatal dexamethasone administration in the infant: long-term follow-up. J Pediatr. 1984 Feb;104(2):259-67. doi: 10.1016/s0022-3476(84)81009-4. PMID 6363659
- [Background] Collaborative Group on Antenatal Steroid Therapy: Prevention of Respiratory Distress Syndrome: Effect of Antenatal Dexamethasone Administration. Hospital and Follow-up Studies. NIH Publication No. 85-2695, 1985.